CLINICAL TRIAL: NCT05147545
Title: Impact of Sport Practice and Hyperlipidic Meal on Free Circulating DNA in Patients With Metastatic Colonic Cancer and Healthy Subjects. Physiological Pilot Study
Brief Title: Impact of Exercise and Hyperlipidic Meal on Free Circulating DNA in Patients With Metastatic Colonic Cancer and Healthy Subjects
Acronym: ASRHACOLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Eurofins Biomnis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP201461; IDRCB 2020-A02872-37 (Other: ANSM); APHP201461 (Other: AP-HP)
Record Dates: First submitted 2021-11-15; First posted 2021-12-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Colon Cancer
Keywords: colon cancer; circulating DNA; Exercise; Meal
MeSH Terms: conditions — Colonic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Physiological pilot study-two groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects free of malignancy (Experimental): Moderate intensity physical effort and meal (once)
  Interventions: Other: Moderate intensity physical effort; Other: Hyperlipidic meal; Diagnostic Test: Measure of circulating DNA
- Patients with colon cancer (Experimental): Low intensity physical effort and meal (visit 1, day of cycle 1 chemotherapy) and low intensity physical effort (visit 2, day of cycle 2 chemotherapy)
  Interventions: Other: Low intensity physical effort; Other: Hyperlipidic meal; Diagnostic Test: Measure of circulating DNA

INTERVENTIONS:
Other: Moderate intensity physical effort — Pedaling 15 minutes at 75 Watt then 100 Watt of the ergometer
  Arms: Subjects free of malignancy
Other: Low intensity physical effort — Pedaling 3 minutes at the 30 Watt level of the ergometer
  Arms: Patients with colon cancer
Other: Hyperlipidic meal — Eating an hyperlipidic meal 60 minutes after a physical effort
Diagnostic Test: Measure of circulating DNA — Multiple measure of circulating DNA: on an empty stomach, at the end of the physical effort, after 15, 30 and 60 minutes of rest, 120 minutes after an hyperlipidic meal.
  An additional measure will occur for subjects free of malignancy during the effort.

SUMMARY:
The study of circulating tumoral DNA makes it possible to study, without invasive procedures or pathological studies, the tumoral DNA circulating in the blood of a patient and its various alterations. In patients with colon-rectal cancer with resected tumor, circulating tumor DNA can be used as a predictive biomarker of metastatic relapse of cancer. However, the routine extension of circulating tumoral DNA remains limited due to several difficulties. One of the pifalls that circulating tumor DNA is greatly diluted by healthy circulating DNA from non-tumor cells. The amount of healthy circulating DNA has been described as being influenced by certain physiological parameters. The aim of the study is to increase knowledge on the influence of physiological factors associated with sports activity and meal on the release kinetics of circulating DNA.

DETAILED DESCRIPTION:
20 subjects free of malignancy (Male-Female Ratio 2 to 1) the variation in the concentration of DNA circulating between the value measured on an empty stomach after 1 hour of rest, then at the end of each of the successive stages of moderate intensity physical effort: pedaling 15 minutes at 75 Watt then 100 Watt of the ergometer. Dosages will be repeated after 15, 30 and 60 minutes of recovery. After an hour of recovery, the subject will be asked to consume a meal rich in fat. The circulating DNA will be measured 2 hours after the end of the meal.

40 patients with colon cancer will be enrolled for a two visit study. The first visit will be planned at the first cycle of chemotherapy, before the chemotherapy. At this visit, the influence of exercise on plasma concentrations of circulating free DNA will also be studied in 40 patients with colon cancer. Free circulating DNA will be measured on an empty stomach after 1 hour of rest, then immediately after low-intensity physical effort : pedaling 3 minutes at the 30 Watt level of the ergometer) and after 15, 30 and 60 minutes of recovery. After an hour of recovery, the subject will be proposed to consume a meal rich in fat. The circulating DNA will be measured 2 hours after the end of the meal. The second visit will be planned at the first second of chemotherapy, before the chemotherapy. Free circulating DNA will be measured on an empty stomach after 1 hour of rest, then immediately after low-intensity physical effort : pedaling 3 min at the 30 Watt level of the ergometer, and after 15, 30 and 60 minutes of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects free of malignancy

   * men or women 40-70 yrs aged
2. Patients with colon cancer

   * men or women 18-85 yrs aged
   * Biopsy-proven colon cancer with indication to chemiotherapy
   * Chemiotherapy (first line or second line) not started

Exclusion Criteria:

1. All subjects

   * Ischemic cardiac history
   * known heart disease
   * blood hemoglobin concentration <8g / dl
   * Acute or chronic systemic illnesses, (apart from diabetes, essential or secondary hypertension for patients)
   * Pregnancy or breastfeeding or in progress
2. Subjects free of malignancy

   * Cardiovascular risk factor (active smoking or greater than 10 pack-years, diabetes, hypertension or known dyslipidemia not controlled by the diet)
   * Glomerular filtration rate estimated by the CKD epi (Chronic Kidney Disease - Epidemiology Collaboration) formula < 60 ml.min-1.1.73 m-²
   * Contraindication to exercise
   * Drug taking in progress (except estrogen-progestogen contraception)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in circulating DNA induced by moderate effort in subjects free of malignacy | 0, 3, 15 minutes of exercise, 15, 30 and 60 minutes of recovery.
  Variation in the concentration of circulating DNA between the value measured after 1 hour of rest, during and at recovery of moderate intensity physical effort

SECONDARY OUTCOMES:
Change in circulating DNA induced by hyperlipidic meal in subjects free of malignacy | 0 minutes (before eating) and 120 minutes after eating
  Variation in the concentration of circulating DNA between the value measured before and after an hyperlipidic meal in subjects free of malignancy
Change in circulating DNA induced by moderate effort in patients with colon cancer | 0, 15, 30 and 60 minutes of recovery.
  Variation in the concentration of circulating DNA between the value measured after 1 hour of rest, during and at recovery of low intensity physical effort
Change in circulating DNA induced by hyperlipidic meal in patients with colon cancer | 0 minutes (before eating) and 120 minutes after eating
  Variation in the concentration of circulating DNA between the value measured before and after an hyperlipidic meal

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LAURENT-PUIG, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris, Hôpital européen Georges Pompidou, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared Supporting Information: Study Protocol Informed Consent Form (ICF)
  Time Frame:
  Two years after the last publication
  Access Criteria:
  Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).